CLINICAL TRIAL: NCT05192252
Title: Correlation Between Seminal Vesicle Size and Duration of Sexual Abstinence
Acronym: AbsVS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: AbsVS
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Suspected Prostate Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The seminal vesicles (SV) are glands that open into the prostatic urethra and secrete seminal fluid, which makes up 50 to 80% of semen. They play an essential role in the male reproductive function. In adults, the size of a seminal vesicle varies from one individual to another. On average, it is 5 to 6 cm long, 1.5 cm wide and 0.5 cm thick. It has a close anatomical relationship with Walsh's vascular-nervous pedicle, which extends the sacro-genital-pubic blades, and is responsible for erection. The reference treatment for localized prostate cancer can consist of two alternatives: either intensity-modulated pelvic radiotherapy with treatment of the entire prostate volume and VS, or surgical removal of the vesiculo-prostatic block in monobloc. It is therefore always extended to the VS.

Magnetic resonance imaging (MRI) is now routinely performed for the initial workup of prostate cancer, with a diagnostic and prognostic role, as invasion of the VS by cancer is recognized as a poor prognostic factor. Some radiology centers recommend 3 days of sexual abstinence to allow a proper seminal vesicle study. Various factors, such as serum testosterone levels, autosomal dominant polycystic kidney disease, smoking, and certain drugs such as SILODOSINE, have been identified as factors that can independently vary seminal vesicle size.

The duration of sexual abstinence since the last ejaculation also appears to be correlated with seminal vesicle volume. Two recent studies found a correlation between the duration of sexual abstinence and seminal vesicle volume measured on MRI in a young population (median age 35.9 and 46.45 years). This population is not superimposable to that of patients managed for prostate cancer whose average age at diagnosis is 70 years.

However, the control and knowledge of the volume of VS, in this specific population, could have an interest in the treatment of prostate cancer:

* In case of pelvic radiotherapy in order to limit the volume of the organ to be irradiated, the toxicity induced to the adjacent organs being directly associated to the delivered dose.
* In case of radical vesiculo-prostatectomy, by surgical way, the lateral dissection of the vasculo-nerveous bands is made more difficult in case of voluminous seminal vesicles with an increased risk of nerve damage.

Investigators hypothesize that the volume of the VS is correlated with the duration of abstinence. Thus, evacuation of seminal fluid by ejaculation at a defined time before curative treatment of prostate cancer, could improve the functional results of pelvic radiotherapy or surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 45 years
* French speaking patient
* Patient performing a prostate MRI for suspected prostate cancer

Exclusion Criteria:

* History of curative treatment for prostate cancer (radical prostatectomy, external radiotherapy, brachytherapy, HIFU, cryotherapy)
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his or her data for this research

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient performing a prostate MRI for suspected prostate cancer, between 07/06/2021 and 30/10/2022.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between seminal vesicle volume measured on MRI and duration of sexual abstinence | Day 1
  This outcome corresponds to the Correlation coefficient between seminal vesicle volume measured on 3 Tesla prostate MRI and duration of sexual abstinence.

CONTACTS AND LOCATIONS:
Overall Officials: Constance MICHEL, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Barrett T, Turkbey B, Choyke PL. PI-RADS version 2: what you need to know. Clin Radiol. 2015 Nov;70(11):1165-76. doi: 10.1016/j.crad.2015.06.093. Epub 2015 Jul 29. PMID 26231470
- [Background] Qi X, Gao XS, Asaumi J, Zhang M, Li HZ, Ma MW, Zhao B, Li FY, Wang D. Optimal contouring of seminal vesicle for definitive radiotherapy of localized prostate cancer: comparison between EORTC prostate cancer radiotherapy guideline, RTOG0815 protocol and actual anatomy. Radiat Oncol. 2014 Dec 20;9:288. doi: 10.1186/s13014-014-0288-1. PMID 25526901
- [Background] Lotti F, Corona G, Vitale P, Maseroli E, Rossi M, Fino MG, Maggi M. Current smoking is associated with lower seminal vesicles and ejaculate volume, despite higher testosterone levels, in male subjects of infertile couples. Hum Reprod. 2015 Mar;30(3):590-602. doi: 10.1093/humrep/deu347. Epub 2015 Jan 6. PMID 25567620
- [Background] Lotti F, Corona G, Maseroli E, Rossi M, Silverii A, Degl'innocenti S, Rastrelli G, Forti G, Maggi M. Clinical implications of measuring prolactin levels in males of infertile couples. Andrology. 2013 Sep;1(5):764-71. doi: 10.1111/j.2047-2927.2013.00114.x. PMID 23970454
- [Background] Bozkurt O, Demir O, Sen V, Esen A. Silodosin causes impaired ejaculation and enlargement of seminal vesicles in sexually active men treated for lower urinary tract symptoms suggestive of benign prostatic hyperplasia. Urology. 2015 May;85(5):1085-1089. doi: 10.1016/j.urology.2015.01.011. Epub 2015 Mar 3. PMID 25744372
- [Background] Joo I, Kim SH, Cho JY. A comparison of seminal vesicle size on CT between autosomal dominant polycystic kidney disease (ADPKD) patients and normal subjects. Acta Radiol. 2010 Jun;51(5):569-72. doi: 10.3109/02841851003652583. PMID 20235741
- [Background] Barrett T, Tanner J, Gill AB, Slough RA, Wason J, Gallagher FA. The longitudinal effect of ejaculation on seminal vesicle fluid volume and whole-prostate ADC as measured on prostate MRI. Eur Radiol. 2017 Dec;27(12):5236-5243. doi: 10.1007/s00330-017-4905-x. Epub 2017 Jul 4. PMID 28677052
- [Background] Yuruk E, Pastuszak AW, Suggs JM 3rd, Colakerol A, Serefoglu EC. The association between seminal vesicle size and duration of abstinence from ejaculation. Andrologia. 2017 Sep;49(7):10.1111/and.12707. doi: 10.1111/and.12707. Epub 2016 Sep 23. PMID 27660049